CLINICAL TRIAL: NCT00430950
Title: Efficacy and Safety of Olmesartan Medoxomil/Hydrochlorothiazide Combination 20/25 mg Versus 40/25 mg in Moderately to Severely Hypertensive Patients Not Adequately Controlled by Olmesartan Medoxomil 40 mg Monotherapy
Brief Title: Combination of Olmesartan and Hydrochlorothiazide in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS866CM-B-E302
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2009-04-20 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2017-10

CONDITIONS: Essential Hypertension
Keywords: Moderate-to-Severe Hypertension; Essential Hypertension; Combination Therapy; Fixed-Combination Dose
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): olmesartan medoximil (OM)/ hydrochlorothiazide (HCTZ) 40/25 mg + OM/HCTZ 20/25 mg matching placebo
  Interventions: Drug: olmesartan medoxomil (OM)+ hydrochlorothiazide (HCTZ) tablets
- 2 (Experimental): olmesartan medoximil (OM)/ hydrochlorothiazide (HCTZ)20/25 mg + OM/HCTZ 40/25 matching placebo
  Interventions: Drug: olmesartan medoxomil (OM)/ hydrochlorothiazide (HCTZ) 20mg/25mg

INTERVENTIONS:
Drug: olmesartan medoxomil (OM)+ hydrochlorothiazide (HCTZ) tablets — olmesartan medoxomil (OM)+ hydrochlorothiazide (HCTZ)tablets 40mg/25mg + 20mg/25mg matching placebo tablets once daily for 8 weeks
  Arms: 1
Drug: olmesartan medoxomil (OM)/ hydrochlorothiazide (HCTZ) 20mg/25mg — olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ)20mg/25mg tablet + 40mg/25mg matching placebo tablet once a day for 8 weeks
  Arms: 2

SUMMARY:
The study will evaluate the blood pressure lowering effects of two different dosages of the combination of olmesartan and hydrochlorothiazide in patients with moderate or severe high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Europeans aged 18 years or older with moderate to severe HTN, defined as follows (conventional BP measurements)

Exclusion Criteria:

* Female patients of childbearing potential pregnant, lactating or planning to become pregnant during the trial period.
* Patients with serious disorders which may limit the ability to evaluate the efficacy or safety of the study medication, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, haematological or oncological, neurological and psychiatric diseases.
* Patients having a history of the following within the last six months:

  * myocardial infarction,
  * unstable angina pectoris,
  * percutaneous coronary intervention,
  * severe heart failure,
  * hypertensive encephalopathy, cerebrovascular accident (stroke) or
  * transient ischaemic attack.
* Patients with clinically significant abnormal laboratory values at screening.
* Patients with secondary HTN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Lars Christian Rump, M.D., Study Chair — University of Ruhr-Bochum
Locations (41):
- Belgium (6):
  - Bruges
  - Brussels
  - Drongen
  - Godinne
  - Mouscron
  - Wetteren
- Germany (14):
  - Berlin
  - Dortmund
  - Essen
  - Frankfurt
  - Goch
  - Hamburg
  - Kallstadt
  - Karlsruhe
  - Kassel
  - Magdeburg
  - Marburg
  - München
  - Wiesbaden
  - Wuppertal
- Netherlands (15):
  - 's-Hertogenbosch
  - Alphen aan den Rijn
  - Amsterdam-Zuidoost
  - Andijk
  - De Bilt
  - Ewijk
  - Heerlen
  - Hengelo
  - Landgraaf
  - Nijmegen
  - Oud-Beijerland
  - Ridderkerk
  - The Hague
  - Wildervank
  - Zwijndrecht
- Slovakia (6):
  - Bratislava
  - Levice
  - Lučenec
  - Nitra
  - Nové Zámky
  - Vráble

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Rosenbaum D, Girerd X. Olmesartan medoxomil combined with hydrochlorothiazide improves 24-hour blood pressure control in moderate-to-severe hypertension. Curr Med Res Opin. 2012 Feb;28(2):179-86. doi: 10.1185/03007995.2011.644626. Epub 2012 Jan 9. PMID 22114906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 92 principal investigators screened patients at clinical sites in Europe (8 in Belgium, 17 in Germany, 12 in the Netherlands, 17 in Poland, 19 in Russia, 10 in Slovakia, and 9 in the Ukraine).Sites were either hospitals or general practitioners.
  First patient in: 05 December 2006 Last patient out: 07 May 2008
Pre-assignment Details: Trial is 2 week taper-off phase and 2 treatment periods. Period I - 8-week open-label OM 40mg. Only non-responders eligible to randomise into Period II. Period II - 8-week double-blind patients assigned into one of two arms. Results provided for Period II only.
Groups:
- OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo: Olmesartan Medoxomil/Hydrochlorothiazide 40/25 mg with 20/25 mg matching placebo
- OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo: Olmesartan Medoxomil/Hydrochlorothiazide 20/25mg + 40/25mg matching placebo
Period: Overall Study
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo
Started | 502 | 508
Completed | 489 | 495
Not Completed | 13 | 13
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — concomitant medication,etc. | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo | Total
Number analyzed (Participants) | 502 | 508 | 1010
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 404 | 422 | 826.0
  >=65 years | 93 | 75 | 168.0
  >= 75 years | 5 (1.0) | 11 (2.2) | 16.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.67) | 54.4 (9.77) | 54.6 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 201 | 395
  Male | 308 | 307 | 615
Race/Ethnicity, Customized [Number; unit: participants]
  European | 502 | 508 | 1010

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Trough Sitting Diastolic Blood Pressure
Description: Change in mean trough sitting diastolic Blood Pressure between OM/HCTZ 20/25 mg vs. 40/25 mg, in those patients inadequately controlled on OM 40 mg monotherapy, after eight weeks of double blind treatment, as compared to baseline.
  Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks
Population: The main analysis will be performed on the full analysis set last observation carried forward (LOCF). Pooling will be applied for small centres.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo
Number analyzed (Participants) | 502 | 508
mm Hg | -11.16 (8.851) | -10.45 (7.928)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; The ANCOVA model included treatment as main effect and baseline mean trough sitting dBP as covariate. Significance level alpha = 5%. Power = 80%. The following statistical superiority hypothesis was tested: Superiority of OM/HCTZ combination therapy 40/25 mg over OM/HCTZ 20/25 mg; Test type: Superiority or Other; p = 0.2648, ANCOVA; Mean Difference (Net) = -0.5, 95% CI [-1.51 to 0.42]

2. Secondary Outcome: Change in Mean Trough Sitting Diastolic Blood Pressure From Week 8(Baseline) to Week 12
Description: Change = Week 12 - Week 8 (baseline).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo
Number analyzed (Participants) | 502 | 508
mm Hg | -9.32 (7.820) | -8.83 (7.584)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.4246, ANCOVA; Mean Difference (Net) = -0.4, 95% CI [-1.26 to 0.53]

3. Secondary Outcome: Change in Sitting Systolic Blood Pressure 4 Weeks and 8 Weeks After Baseline.
Description: 4 weeks Change = Week 12 - Week 8 (baseline). 8 weeks Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo
Number analyzed (Participants) | 502 | 508
mm Hg
  Change from baseline (Week 8) to Week 16 in sBP | -17.41 (13.930) | -17.09 (13.126)
  Change from baseline (Week 8) to Week 12 in sBP | -14.07 (12.654) | -13.80 (12.519)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.7019, ANCOVA; Mean Difference (Net) = -0.3, 95% CI [-1.84 to 1.24] — refers to 8 week change; from week 8 to week 16
Statistical Analysis 2: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.7328, ANCOVA; Mean Difference (Net) = -0.3, 95% CI [-1.71 to 1.21] — refers to 4 week change; from week 8 to week 12

4. Secondary Outcome: Change in Daytime, Nighttime and 24-hour Blood Pressure Evaluated by Ambulatory Blood Pressure Monitoring 8 Weeks After Baseline.
Description: Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks
Population: Exploratory analysis: ANCOVA was used to compare the differences in change from baseline (Visit 4, Week 8) to Week 16 (Visit 6) in daytime, nighttime and 24-hr ABPM dBP and sBP.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo
Number analyzed (Participants) | 442 | 442
mm Hg
  Change from Week 8 to Wk 16 in mean 24-hr ABPM dBP | -9.2 (8.69) | -7.6 (8.03)
  Change from Week 8 to wk16 in daytime ABPM dBP | -9.3 (9.18) | -7.7 (8.48)
  Change from Week 8 to wk16 in nighttime ABPM dBP | -8.6 (9.52) | -7.0 (9.49)
  Change from Week 8 to wk16 in mean 24-hr ABPM sBP | -14.7 (13.75) | -12.0 (11.81)
  Change from Week 8 to wk16 in daytime ABPM sBP | -15.0 (14.36) | -12.3 (12.45)
  Change from Week 8 to wk16 in nighttime ABPM sBP | -13.4 (14.59) | -10.7 (13.16)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.0016, ANCOVA; Mean Difference (Net) = -1.6, 95% CI [-2.58 to -0.60] — 24 hour Ambulatory Blood Pressure Monitoring (ABPM) diastolic blood pressure (dBP)
Statistical Analysis 2: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.0031, ANCOVA; Mean Difference (Net) = -1.6, 95% CI [-2.61 to -0.53] — daytime Ambulatory Blood Pressure Monitoring (ABPM) diastolic blood pressure (dBP)
Statistical Analysis 3: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.0073, ANCOVA; Mean Difference (Net) = -1.5, 95% CI [-2.58 to -0.40] — night-time Ambulatory Blood Pressure Monitoring (ABPM) diastolic blood pressure (dBP)
Statistical Analysis 4: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.0021, ANCOVA; Mean Difference (Net) = -2.3, 95% CI [-3.71 to -0.82] — 24 hour Ambulatory Blood Pressure Monitoring (ABPM) systolic blood pressure (sBP)
Statistical Analysis 5: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.0031, ANCOVA; Mean Difference (Net) = -2.3, 95% CI [-3.76 to -0.76] — daytime Ambulatory Blood Pressure Monitoring (ABPM) systolic blood pressure (sBP)
Statistical Analysis 6: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; p = 0.0104, ANCOVA; Mean Difference (Net) = -2.0, 95% CI [-3.61 to -0.48] — night-time Ambulatory Blood Pressure Monitoring (ABPM) systolic blood pressure (sBP)

5. Secondary Outcome: Number of Participants Achieving Blood Pressure Goal.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo | OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo
Number analyzed (Participants) | 502 | 508
participants | 260 | 255
Statistical Analysis 1: Comparison: OM/HCTZ 40/25 mg + 20/25 mg Matching Placebo vs OM/HCTZ 20/25 mg + 40/25 mg Matching Placebo; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI [0.85 to 1.40]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of Study shall not be published without prior express written consent and approval of Sponsor. If Contractor wishes to use data generated at Sites by Investigator, such data includes but not limited to data used in collection of metrics, copy of any intended publication, details of use must be sent in writing to Quintiles and Sponsor for review. Sponsor has right to change proposed publication and/or prohibit publication and Contractor must comply with requirements of Sponsor